CLINICAL TRIAL: NCT04309110
Title: Evaluation of the Adhesive Strength of the Geko™ X-T3 Neuromuscular Stimulator Incorporating a New Skin Adhesive Hydrogel Formulation Designated KM40C
Brief Title: Efficacy of Adhesive Strength of New Hydrogel Formulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Firstkind Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: FSK-R&D-001
Record Dates: First submitted 2020-03-12; First posted 2020-03-16 (Actual); Results first posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2023-07

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: A prospective, non-blinded service evaluation of two sequential groups of patients carried out in two phases.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care with geko™ T3 device (No Intervention): Current geko™ device incorporating hydrogel adhesive designated KM10T
- geko™ X-T3 (Active Comparator): Next generation geko™ device incorporating new hydrogel adhesive designated KM40C
  Interventions: Device: or geko™ X-T3

INTERVENTIONS:
Device: or geko™ X-T3 — The geko™ X-T3 is a next generation self adhesive medical device incorporating a new formulation skin adhesive. It is about the size of a wrist watch which attaches to the side of the knee and when switched on, gentle painless electrical pulses are produced which contract the calf muscles and increase blood flow to the lower leg. The only difference between the currently used geko™ T3 device and the new geko™ XT-3 device is the adhesive used to attach each device to the skin.
  Arms: geko™ X-T3

SUMMARY:
The study will look at the stickiness of a new skin adhesive incorporated into a new next generation geko™ device called the geko™ X-T3 and compare it to the adhesive currently used into the geko™ T3 device. The study is for people who are in hospital in the Acute Stroke Unit, and who will be receiving daily treatment with the geko™ T3 device in line with UK guidelines as part of their standard acute stroke care and venous thromboembolism prevention.

DETAILED DESCRIPTION:
The new skin adhesive incorporated into the next generation geko™ device designated geko™ XT-3 has previously been tested to current international biocompatibility standards (ISO10993) , however the skin adhesive strength of the geko™ X-T3 device compared to that of the current geko™ T3 device has not yet been tested. The reason behind the study is to compare the skin adhesive strength of the two devices in a similar use environment, to determine whether the geko™ XT-3 device will be a suitable replacement for the geko™ T3 device.

In total 40 people who are patients in hospital in the Acute Stroke Unit, and who will receive daily treatment with the geko™ T3 device as part of their acute stroke care and venous thromboembolism prevention pathway will be asked if they would like to take part in the study. 20 patients will receive their normal daily treatment with the currently in use geko™ T3 device and 20 patients will receive their normal daily treatment with the new geko™ XT-3 device which has the new skin adhesive.

Phase 1 will take place before Phase 2 and each phase will last for a maximum of 10 days or until patients are able to walk independently. Each day during the study and after their standard treatment has been completed, a member of the healthcare team will ask the patient questions about their experience with geko™ device and the answers recorded.

The standard acute stroke care patients receive when on the study will not be affected, regardless of which geko™ device they receive and because the study fits into the normal treatment given to these stroke patients whilst in hospital there will be no additional study visits.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥ 18 years
* Currently an in-patient hospitalised for acute stroke
* Use of geko™ as a mechanical prophylaxis strategy for venous thromboembolism
* Patient understands and is willing to participate in the study and is able to comply with study procedures

Exclusion Criteria:

* Pregnancy or breast feeding
* Use of any neuro-modulation device other than geko™
* Participation in any other clinical study that may interfere with the outcome of either study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-07-13 (Actual); Primary Completion 2021-11-25 (Actual); Study Completion 2021-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Indira Natarajan, FRCP, Principal Investigator — University Hospitals of North Midlands NHS Trust
Locations (1):
- University Hospitals of North Midlands NHS Trust, Stoke-on-Trent, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Device official website — http://www.gekodevices.com/en-uk/

RESULTS

PARTICIPANT FLOW:
Groups:
- Geko™ T3 Device: Current geko™ device incorporating hydrogel adhesive designated KM10T
- Geko™ X-T3 Device: Next generation geko™ device incorporating new hydrogel adhesive designated KM40C
Period: Overall Study
Arm/Group | Geko™ T3 Device | Geko™ X-T3 Device
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Geko™ T3 Device | Geko™ X-T3 Device | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Customized [Count of Participants; unit: Participants]
  41-50 | 0 | 3 | 3
  51-60 | 4 | 6 | 10
  61-70 | 4 | 2 | 6
  71-80 | 7 | 7 | 14
  >81 | 5 | 2 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 13 | 11 | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of the Skin Adhesive Strength of Hydrogel KM40C Compared to That of Hydrogel KM10T.
Description: Self reported - how well did the geko™ device stick to the patients leg? Scale 1-5, Lowest score indicates best adhesion.
Time Frame: 10 days
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Geko™ T3 Device | Geko™ X-T3 Device
Number analyzed (Participants) | 20 | 20
score on a scale | 1.52 (0.10) | 1.23 (0.05)

2. Secondary Outcome: Incidence of Adverse Events
Description: Reporting of the incidence of adverse events , incidence of serious adverse events, incidence of study treatment related adverse events, and the incidence of device related adverse events
Time Frame: 10 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Maximum of 10 days from trial inclusion
Arm/Group | Geko™ T3 Device | Geko™ X-T3 Device
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 1/20 | 1/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Geko™ T3 Device (N=20) | Geko™ X-T3 Device (N=20)
Rash at site of geko™ device application (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-29): https://cdn.clinicaltrials.gov/large-docs/10/NCT04309110/Prot_SAP_000.pdf